CLINICAL TRIAL: NCT00521976
Title: An Investigation of Activated Factor XII (Fxlla) as a Prognostic Marker.
Brief Title: Risk Markers in the Acute Coronary Syndromes
Acronym: RACS
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Helse Vest (Other); Axis-Shield, Dundee, UK (Unknown)
Responsible Party: Sponsor
Other Study IDs: NSD9253
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Results first posted 2009-08-11 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2015-05

CONDITIONS: Chest Pain; Coronary Artery Disease; Unstable Angina Pectoris; Myocardial Infarction
Keywords: Risk assessment; Chest pain; Coronary Artery Disease; Acute coronary syndromes; Factor XIIa; B-type natriuretic peptide (BNP); high-sensitive C-reactive protein (hsCRP); Omega-3
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease; Angina, Unstable; Myocardial Infarction; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Citrated plasma, EDTA-plasma and packed red blood cells are kept in suitable aliquots at -80 degrees Celcius.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chest pain: Men and women admitted with chest pain and suspected acute coronary syndrome (ACS).

SUMMARY:
The main aim of this trial is to assess the long-term prognostic value of different types of Factor XIIa in an unselected, single center series of 871 chest pain patients admitted to the emergency unit, employing blood samples collected at admission.

The second purpose of this study is to assess the incremental prognostic value of B-type natriuretic peptide (BNP) and high-sensitive C-reactive protein (hsCRP).

A third purpose of this study is to evaluate the prognostic impact of the Omega-3 Index which is a measure of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) relative to other fatty acids in the erythrocyte membrane.

DETAILED DESCRIPTION:
BACKGROUND Cardiac troponins are sensitive markers for myocardial injury in ACS and even a minor elevation of cardiac troponins is associated with an increased risk for future adverse coronary events. However, a detectable troponin release occurs only in a part of patients admitted with ACS. The clinical outcomes and further prognosis of patients with ACS with absent TnT release vary widely, and the identification of potential high-risk patients with troponin negative ACS still remains a major problem in clinical routine. Therefore, the aim of this study is focused on identifying new biomarkers for risk stratification.

Activated Factor XII: Activated Factor XII leads to contact activation and a number of pathophysiological processes, including hypotension, inflammation, thrombosis and fibrinolysis, are affected by contact activation following the activation of XIIa. Several studies have demonstrated a relation between XIIa and coronary artery heart disease (CAD) (1,2,3,4) and that XIIa levels post MI predict recurrent coronary occlusive events and play a role as an independent risk marker in these patients (5).

However, the detailed mechanisms of XIIa's actions in CAD still remain uncertain although recent findings in animal studies using FXII deficient mice indicate that Factor XII is essential for arterial thrombus formation (6).

Recent research indicates that in-vivo XIIa exists in multiple types and that in-vivo XIIa can exist in the circulation complexed to a variety of other proteins (7). To date, no data exist on the prognostic value of specific in-vivo types of XIIa on outcome in patients with chest pain and/or ACS.

B-type natriuretic peptide: B-type natriuretic peptide (BNP) is a counter-regulatory peptide hormone predominantly synthesized in the ventricular myocardium. BNP is released into the circulation in response to ventricular dilatation and pressure overload, and reflects ventricular wall stress and tissue hypoxia rather than cell injury per se (8, 9). It is a well known marker of left ventricular dysfunction and heart failure (HF), and it provides prognostic information beyond and above left ventricular ejection fraction (LVEF) in patients with an acute coronary syndrome (ACS) (10). This marker of neurohormonal activation and inflammation plays a pivotal role across the spectrum of ACS, including patients with ST-elevation myocardial infarction (MI) and non ST-elevation ACS (NSTE-ACS). Previous studies have demonstrated that BNP measured in the first days after the onset of symptoms independently predicts mortality, HF, and new MI in this patient population. Elevated natriuretic peptides at presentation have been shown to identify patients with ACS who are at higher risk of death and HF, and it adds information to that provided by the troponins (11-13). However, in a low-risk population the association between elevated BNP and survival is attenuated when adjustment is made for echocardiographic variables (in addition to clinical covariates), as shown by Wang and colleagues. In addition, they did not find any association between baseline BNP and the risk of coronary heart disease (CHD) (14).

High-sensitive C-reactive protein (hsCRP): C-reactive protein (CRP) is an acute-phase reactant that is produced in response to acute injury, infection or other inflammation stimuli. It is a marker for underlying systemic inflammation and plays an important role in the initiation and propagation of atherosclerosis and ultimately to plaque rupture and the ensuing thrombotic complication (15) Elevated levels of CRP were first reported in patients hospitalized with NSTE-ACS in the early 1990s (16, 17). Through the use of appropriate high-sensitive assays, it has been possible to investigate the relationship between plasma CRP levels that previously were considered to be normal and cardiovascular disease (CVD). Nevertheless, it is still under debate which markers should be preferred for risk prediction (18, 19). It has been suggested that the combined evaluation of BNP and CRP may yield incremental prognostic information in the risk stratification of patients with ACS (20), and their combined use has been shown to improve long-term risk prediction of mortality in patients with stable CHD (21). To our knowledge, there are limited data available that directly compare these two markers in a prospective manner in an unselected patient population presenting to the emergency department (ED) with chest pain. In addition, their role in risk stratification in patients with ACS is still under evaluation, and therefore additional investigations are necessary.

Omega- 3 Index: The value of the Omega-3 Index as a prognostic marker in the acute coronary syndromes is still under investigation.

STUDY DESIGN This prospective single center observational non-invasive trial includes 871 men and women admitted with chest pain and potential ACS at the Stavanger University Hospital between November 2002 and October 2003. Blood samples were collected immediately following admission. Patients were stratified according to peak troponin T (TnT) release following admission; i.e. 1) patients with an admission TnT exceeding 0.05 ng/mL, and 2) patients with a peak TnT level of 0.05 ng/mL or lower.

Assessment of a history of previous MI, angina pectoris (AP), congestive heart failure (CHF), diabetes mellitus and arterial hypertension was based on hospital records and personal interview. Electrocardiographic findings at admission were classified according to the presence of ST segment changes.

Written informed consent was obtained from all patients. Survival status, date and cause of death and clinical data were obtained by telephone interview and hospital journal reports at 4 predefined time points (30 days, 6, 12 and 24 months) during the two year follow-up period. In case of incapacity to provide information, the general practitioner or nursery home were contacted for relevant data. Hospital journals were searched for confirmation of reported data.

Primary Outcome Measures:

* During follow-up
* All cause death
* Non-fatal acute myocardial infarction (MI)
* Combined endpoint of all cause death or non-fatal acute MI
* Combined endpoint of cardiovascular death or non-fatal acute MI

Secondary Outcome Measures:

* During follow-up
* Acute hospitalizations for angina
* Myocardial revascularization

STEERING COMMITTEE

* Professor Dennis WT Nilsen MD PhD, Department of Heart Disease, Stavanger University Hospital
* Heidi Grundt MD PhD Department of Medicine, Stavanger University Hospital
* Øyvind Hetland MD PhD, Department of Clinical Chemistry, Stavanger University Hospital
* Ole Kristensen MD, Department of Clinical Chemistry, Stavanger University Hospital

BIOLOGICAL SAMPLE OWNERSHIP. The biological samples are owned by Stavanger University Hospital and their use for scientific purposes is administered by the Steering Committee.

DATA OWNERSHIP AND PUBLICATION OF RESULTS. The RACS Steering Committee has the ownership of all data registered in the RACS database, and any use of these data including the preparation and publication of scientific reports must be approved by the Steering Committee. Scientific articles will be published by RACS investigators or by authors mentioned by name. The author sequence should be approved by the Steering Committee and based upon contribution. Incentives to involve articles as part of a doctoral thesis should be encouraged. All collaborators in the study will be mentioned by name in an Appendix section of the main article from the study. The results will be published in peer-reviewed scientific journals and in magazines for the general public.

ELIGIBILITY:
Inclusion Criteria:

* adults > 18 years able to give informed consent
* a history of chest pain or other symptoms suggestive of an ACS leading to admission at the emergency unit

Exclusion Criteria:

* < 18 years of age
* Unwillingness or incapacity to provide informed consent
* Prior admission resulting in inclusion in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 871 men and women admitted with chest pain and potential acute cornary syndrome (ACS) at the Stavanger University Hospital between November 2002 and October 2003.
Sampling Method: Probability Sample
Enrollment: 871 (Actual)
Dates: Start 2002-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis WT Nilsen, MD PhD FESC, Principal Investigator — Stavanger University Hospital, Dept. of Cardiology
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway

REFERENCES:
- [Background] Miller GJ, Esnouf MP, Burgess AI, Cooper JA, Mitchell JP. Risk of coronary heart disease and activation of factor XII in middle-aged men. Arterioscler Thromb Vasc Biol. 1997 Oct;17(10):2103-6. doi: 10.1161/01.atv.17.10.2103. PMID 9351378
- [Background] Zito F, Drummond F, Bujac SR, Esnouf MP, Morrissey JH, Humphries SE, Miller GJ. Epidemiological and genetic associations of activated factor XII concentration with factor VII activity, fibrinopeptide A concentration, and risk of coronary heart disease in men. Circulation. 2000 Oct 24;102(17):2058-62. doi: 10.1161/01.cir.102.17.2058. PMID 11044420
- [Background] Cooper JA, Miller GJ, Bauer KA, Morrissey JH, Meade TW, Howarth DJ, Barzegar S, Mitchell JP, Rosenberg RD. Comparison of novel hemostatic factors and conventional risk factors for prediction of coronary heart disease. Circulation. 2000 Dec 5;102(23):2816-22. doi: 10.1161/01.cir.102.23.2816. PMID 11104738
- [Background] Kohler HP, Carter AM, Stickland MH, Grant PJ. Levels of activated FXII in survivors of myocardial infarction--association with circulating risk factors and extent of coronary artery disease. Thromb Haemost. 1998 Jan;79(1):14-8. PMID 9459314
- [Background] Pritchard D, Polwart R. In-vivo, activated factor XII exists in multiple forms, but predominantly as a 53 kD Species. J Thromb and Haemost 2005; Suppl.1; ISSN 1740-3340.
- [Background] Maeda K, Tsutamoto T, Wada A, Hisanaga T, Kinoshita M. Plasma brain natriuretic peptide as a biochemical marker of high left ventricular end-diastolic pressure in patients with symptomatic left ventricular dysfunction. Am Heart J. 1998 May;135(5 Pt 1):825-32. doi: 10.1016/s0002-8703(98)70041-9. PMID 9588412
- [Background] Nakagawa O, Ogawa Y, Itoh H, Suga S, Komatsu Y, Kishimoto I, Nishino K, Yoshimasa T, Nakao K. Rapid transcriptional activation and early mRNA turnover of brain natriuretic peptide in cardiocyte hypertrophy. Evidence for brain natriuretic peptide as an "emergency" cardiac hormone against ventricular overload. J Clin Invest. 1995 Sep;96(3):1280-7. doi: 10.1172/JCI118162. PMID 7657802
- [Background] Richards AM, Nicholls MG, Espiner EA, Lainchbury JG, Troughton RW, Elliott J, Frampton C, Turner J, Crozier IG, Yandle TG. B-type natriuretic peptides and ejection fraction for prognosis after myocardial infarction. Circulation. 2003 Jun 10;107(22):2786-92. doi: 10.1161/01.CIR.0000070953.76250.B9. Epub 2003 May 27. PMID 12771003
- [Background] de Lemos JA, Morrow DA, Bentley JH, Omland T, Sabatine MS, McCabe CH, Hall C, Cannon CP, Braunwald E. The prognostic value of B-type natriuretic peptide in patients with acute coronary syndromes. N Engl J Med. 2001 Oct 4;345(14):1014-21. doi: 10.1056/NEJMoa011053. PMID 11586953
- [Background] Morrow DA, de Lemos JA, Sabatine MS, Murphy SA, Demopoulos LA, DiBattiste PM, McCabe CH, Gibson CM, Cannon CP, Braunwald E. Evaluation of B-type natriuretic peptide for risk assessment in unstable angina/non-ST-elevation myocardial infarction: B-type natriuretic peptide and prognosis in TACTICS-TIMI 18. J Am Coll Cardiol. 2003 Apr 16;41(8):1264-72. doi: 10.1016/s0735-1097(03)00168-2. PMID 12706919
- [Background] Omland T, Persson A, Ng L, O'Brien R, Karlsson T, Herlitz J, Hartford M, Caidahl K. N-terminal pro-B-type natriuretic peptide and long-term mortality in acute coronary syndromes. Circulation. 2002 Dec 3;106(23):2913-8. doi: 10.1161/01.cir.0000041661.63285.ae. PMID 12460871
- [Background] Wang TJ, Larson MG, Levy D, Benjamin EJ, Leip EP, Omland T, Wolf PA, Vasan RS. Plasma natriuretic peptide levels and the risk of cardiovascular events and death. N Engl J Med. 2004 Feb 12;350(7):655-63. doi: 10.1056/NEJMoa031994. PMID 14960742
- [Background] Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26. doi: 10.1056/NEJM199901143400207. No abstract available. PMID 9887164
- [Background] Liuzzo G, Biasucci LM, Gallimore JR, Grillo RL, Rebuzzi AG, Pepys MB, Maseri A. The prognostic value of C-reactive protein and serum amyloid a protein in severe unstable angina. N Engl J Med. 1994 Aug 18;331(7):417-24. doi: 10.1056/NEJM199408183310701. PMID 7880233
- [Background] Berk BC, Weintraub WS, Alexander RW. Elevation of C-reactive protein in "active" coronary artery disease. Am J Cardiol. 1990 Jan 15;65(3):168-72. doi: 10.1016/0002-9149(90)90079-g. PMID 2296885
- [Background] de Lemos JA. The latest and greatest new biomarkers: which ones should we measure for risk prediction in our practice? Arch Intern Med. 2006 Dec 11-25;166(22):2428-30. doi: 10.1001/archinte.166.22.2428. No abstract available. PMID 17159006
- [Background] Rothenbacher D, Koenig W, Brenner H. Comparison of N-terminal pro-B-natriuretic peptide, C-reactive protein, and creatinine clearance for prognosis in patients with known coronary heart disease. Arch Intern Med. 2006 Dec 11-25;166(22):2455-60. doi: 10.1001/archinte.166.22.2455. PMID 17159010
- [Background] Kim H, Yang DH, Park Y, Han J, Lee H, Kang H, Park HS, Cho Y, Chae SC, Jun JE, Park WH. Incremental prognostic value of C-reactive protein and N-terminal proB-type natriuretic peptide in acute coronary syndrome. Circ J. 2006 Nov;70(11):1379-84. doi: 10.1253/circj.70.1379. PMID 17062957
- [Background] Ndrepepa G, Kastrati A, Braun S, Mehilli J, Niemoller K, von Beckerath N, von Beckerath O, Vogt W, Schomig A. N-terminal probrain natriuretic peptide and C-reactive protein in stable coronary heart disease. Am J Med. 2006 Apr;119(4):355.e1-8. doi: 10.1016/j.amjmed.2005.10.060. PMID 16564781
- [Background] Harris WS, Sands SA, Windsor SL, Ali HA, Stevens TL, Magalski A, Porter CB, Borkon AM. Omega-3 fatty acids in cardiac biopsies from heart transplantation patients: correlation with erythrocytes and response to supplementation. Circulation. 2004 Sep 21;110(12):1645-9. doi: 10.1161/01.CIR.0000142292.10048.B2. Epub 2004 Sep 7. PMID 15353491
- [Result] Ponitz V, Pritchard D, Grundt H, Nilsen DW. Specific types of activated Factor XII increase following thrombolytic therapy with tenecteplase. J Thromb Thrombolysis. 2006 Dec;22(3):199-203. doi: 10.1007/s11239-006-9031-6. PMID 17111198
- [Result] Ponitz V, Pritchard D, Grundt H, Mehus MB, Nilsen DW. Changes of plasma activated Factor XII type A (XIIaA) concentrations following percutaneous coronary intervention (PCI). J Thromb Thrombolysis. 2007 Oct;24(2):131-5. doi: 10.1007/s11239-007-0041-9. Epub 2007 May 11. PMID 17492403
- [Result] Brugger-Andersen T, Hetland O, Ponitz V, Grundt H, Nilsen DW. The effect of primary percutaneous coronary intervention as compared to tenecteplase on myeloperoxidase, pregnancy-associated plasma protein A, soluble fibrin and D-dimer in acute myocardial infarction. Thromb Res. 2007;119(4):415-21. doi: 10.1016/j.thromres.2006.03.009. Epub 2006 May 2. PMID 16650886
- [Result] Ponitz V, Brugger-Andersen T, Pritchard D, Grundt H, Staines H, Nilsen DW; RACS Study Group. Activated factor XII type A predicts long-term mortality in patients admitted with chest pain. J Thromb Haemost. 2009 Feb;7(2):277-87. doi: 10.1111/j.1538-7836.2008.03248.x. Epub 2008 Dec 1. PMID 19054318
- [Result] Brugger-Andersen T, Ponitz V, Staines H, Grundt H, Hetland O, Nilsen DW. The prognostic utility of D-dimer and fibrin monomer at long-term follow-up after hospitalization with coronary chest pain. Blood Coagul Fibrinolysis. 2008 Oct;19(7):701-7. doi: 10.1097/MBC.0b013e32830b1512. PMID 18832914
- [Result] Brugger-Andersen T, Ponitz V, Staines H, Pritchard D, Grundt H, Nilsen DW. B-type natriuretic peptide is a long-term predictor of all-cause mortality, whereas high-sensitive C-reactive protein predicts recurrent short-term troponin T positive cardiac events in chest pain patients: a prognostic study. BMC Cardiovasc Disord. 2008 Nov 25;8:34. doi: 10.1186/1471-2261-8-34. PMID 19032759
- [Result] Aarsetoy H, Ponitz V, Nilsen OB, Grundt H, Harris WS, Nilsen DW. Low levels of cellular omega-3 increase the risk of ventricular fibrillation during the acute ischaemic phase of a myocardial infarction. Resuscitation. 2008 Sep;78(3):258-64. doi: 10.1016/j.resuscitation.2008.04.007. Epub 2008 Jun 16. PMID 18556107
- [Result] Aarsetoey H, Ponitz V, Grundt H, Staines H, Harris WS, Nilsen DW. (n-3) Fatty acid content of red blood cells does not predict risk of future cardiovascular events following an acute coronary syndrome. J Nutr. 2009 Mar;139(3):507-13. doi: 10.3945/jn.108.096446. Epub 2009 Jan 21. PMID 19158216
- [Result] Naesgaard PA, Ponitz V, Aarsetoey H, Brugger-Andersen T, Grundt H, Harris WS, Staines H, Nilsen DW. Prognostic utility of vitamin D in acute coronary syndrome patients in coastal Norway. Dis Markers. 2015;2015:283178. doi: 10.1155/2015/283178. Epub 2015 Feb 5. PMID 25722531
- [Result] Mjelva OR, Brugger-Andersen T, Ponitz V, Grundt H, Kontny F, Staines H, Nilsen DW. Long-term prognostic utility of PAPP-A and calprotectin in suspected acute coronary syndrome. Scand Cardiovasc J. 2013 Apr;47(2):88-97. doi: 10.3109/14017431.2013.764571. Epub 2013 Feb 13. PMID 23406538
- [Derived] Nilsen DWT, Aarsetoey H, Poenitz V, Brugger-Andersen T, Harris WS, Staines H, Grundt H. Dihomo-gamma-linolenic acid (DGLA) is inversely related to risk for cardiac death and cardiovascular events during 2 years follow-up after admission for an acute coronary syndrome. Prostaglandins Leukot Essent Fatty Acids. 2025 Jul;205:102684. doi: 10.1016/j.plefa.2025.102684. Epub 2025 Apr 10. PMID 40245567
- [Derived] Andersen T, Ueland T, Aukrust P, Nilsen DWT, Grundt H, Staines H, Ponitz V, Kontny F. Procollagen type 1 N-terminal propeptide is associated with adverse outcome in acute chest pain of suspected coronary origin. Front Cardiovasc Med. 2023 Sep 4;10:1191055. doi: 10.3389/fcvm.2023.1191055. eCollection 2023. PMID 37731526
- [Derived] Andersen T, Ueland T, Aukrust P, Nilsen DW, Grundt H, Staines H, Kontny F. Podocan and Adverse Clinical Outcome in Patients Admitted With Suspected Acute Coronary Syndromes. Front Cardiovasc Med. 2022 May 20;9:867944. doi: 10.3389/fcvm.2022.867944. eCollection 2022. PMID 35669474
- [Derived] Aarsetoy R, Ueland T, Aukrust P, Michelsen AE, Leon de la Fuente R, Grundt H, Staines H, Nygaard O, Nilsen DWT. Complement component 7 is associated with total- and cardiac death in chest-pain patients with suspected acute coronary syndrome. BMC Cardiovasc Disord. 2021 Oct 14;21(1):496. doi: 10.1186/s12872-021-02306-w. PMID 34649504
- [Derived] Aarsetoy R, Ueland T, Aukrust P, Michelsen AE, de la Fuente RL, Ponitz V, Brugger-Andersen T, Grundt H, Staines H, Nilsen DWT. Angiopoietin-2 and angiopoietin-like 4 protein provide prognostic information in patients with suspected acute coronary syndrome. J Intern Med. 2021 Oct;290(4):894-909. doi: 10.1111/joim.13339. Epub 2021 Jul 8. PMID 34237166
- [Derived] Ponitz V, Brugger-Andersen T, Pritchard D, Grundt H, Staines H, Nilsen DW; RACS study group. Activated factor XII type A and B-type natriuretic peptide are complementary and incremental predictors of mortality in patients following admission with acute coronary syndrome. Blood Coagul Fibrinolysis. 2009 Dec;20(8):652-60. doi: 10.1097/MBC.0b013e32832fa814. PMID 19809305
- [Derived] Brugger-Andersen T, Ponitz V, Kontny F, Staines H, Grundt H, Sagara M, Nilsen DW. The long pentraxin 3 (PTX3): a novel prognostic inflammatory marker for mortality in acute chest pain. Thromb Haemost. 2009 Sep;102(3):555-63. doi: 10.1160/TH09-02-0137. PMID 19718477

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive recruitment at Stavanger University Hospital.
Groups:
- Group 1: Men and women admitted with chest pain and a suspicious acute coronary syndrome (ACS)
Period: Overall Study
Arm/Group | Group 1
Started | 871
Completed | 871
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 871
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 300
  >=65 years | 571
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 340
  Male | 531
Region of Enrollment [Number; unit: participants]
  Norway | 871

OUTCOME MEASURES:

1. Primary Outcome: Total Mortality.
Time Frame: 24 months.
Measure: Number; unit: Participants.
Arm/Group | Group 1
Number analyzed (Participants) | 871
Participants. | 138

2. Secondary Outcome: Recurrent Troponin-T (TnT) Positive Events
Description: Recurrent Troponin-T (TnT) positive events; Symptoms of coronary ischemia associated with TnT >0.05 ng/mL with a pattern of gradual rise and fall in TnT
Time Frame: 24 months.
Measure: Number; unit: Participants
Arm/Group | Group 1
Number analyzed (Participants) | 871
Participants | 155

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/871
Other Adverse Events (participants affected / at risk) | 0/871

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less